CLINICAL TRIAL: NCT06330168
Title: The Analgesic Value of Paravertebral Calcitonin in Patients Undergoing Thoracotomy
Brief Title: Paravertebral Calcitonin in Thoracotomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, lecturer of anesthesiology, surgical intensive care and pain medicine Tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 36264PR573/2/24
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Calcitonin; Paravertebral; Thoracotomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine-calcitonin-fentanyl group (Experimental): thoracic paravertebral block using 20 mL 0.25% bupivacaine, 100 micrograms of fentanyl (2ml), and 100 IU of calcitonin (1ml)
  Interventions: Drug: bupivacaine-calcitonin-fentanyl
- bupivacaine-fentanyl group (Placebo Comparator): thoracic paravertebral block using 20 mL 0.25% bupivacaine, 100 micrograms of fentanyl (2ml), and 1 ml saline 0.9%.
  Interventions: Drug: Bupivacaine-fentanyl

INTERVENTIONS:
Drug: bupivacaine-calcitonin-fentanyl — pre-induction single shot thoracic paravertebral block using 20 mL 0.25% bupivacaine, 100 micrograms of fentanyl (2ml), and 100 IU of calcitonin (1ml).
  Arms: bupivacaine-calcitonin-fentanyl group
Drug: Bupivacaine-fentanyl — pre-induction single shot thoracic paravertebral block using 20 mL 0.25% bupivacaine, 100 micrograms of fentanyl (2ml), and 1 ml saline 0.9%.
  Arms: bupivacaine-fentanyl group

SUMMARY:
This prospective randomized double-blinded controlled study will be conducted to evaluate the effect of adding calcitonin to bupivacaine in thoracic paravertebral block for patients undergoing thoracotomy.

DETAILED DESCRIPTION:
Single-shot thoracic paravertebral block combined with intravenous analgesia is one of the regional techniques used for controlling pain in patients undergoing thoracic surgery. However, few articles demonstrated its effects on acute pain and chronic pain after thoracotomy and revealed high postoperative opioid consumption and inability to reduce the incidence of chronic pain.

Calcitonin has previously been shown to be effective in the management of acute pain following amputation, vertebral fractures and other neuropathic conditions.

Using calcitonin as an additive in thoracic paravertebral block was not evaluated in previous studies, investigators conducted this study based on the hypothesis that calcitonin use as an additive in thoracic paravertebral block for patients undergoing thoracotomy may have extended analgesic effects regarding decreasing postoperative pain scores, opioid consumption, and this value may decrease the incidence of chronic post-thoracotomy pain.

In both groups, ultrasound-guided thoracic paravertebral block will be performed before anesthetic induction using a high-frequency linear probe after identifying the paravertebral space of the proposed level of intercostal skin incision.General anesthesia in both groups will be similar.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* American society of anesthesiology (ASA) physical status of I-III
* scheduled for elective thoracotomy

Exclusion Criteria:

* Contraindication to thoracic paravertebral block as coagulopathy or local anesthetic allergy.
* Pregnancy
* History of cardiovascular and gastro-esophageal surgery
* Preexisting pain syndrome or psychological disorders
* Severe hepatic, cardiovascular, or renal disorders
* Allergy to calcitonin
* Patients who will be re-operated and who will report infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | from the end of surgery until the end of the first postoperative day
  Total morphine dose consumed in the first 24 hour after surgery
Incidence of chronic pain at 3 months after surgery | 3 months after surgery
  chronic pain at 3 months after surgery

SECONDARY OUTCOMES:
numerical rating scale scores | from arrival to the post-anesthesia care unit until 48 hour after surgery.
  A 0-10 numerical rating scale ( 0 means no pain and 10 means the worst pain) at coughing and at rest will be assessed by an investigator during the first and second day post operation
incidence of chronic pain | 12 months after surgery
  chronic pain at 6, 9, and 12 months after surgery
Side effects | first postoperative day
  hypotension, postoperative nausea and vomiting
Intensity of chronic pain | 12 months after surgery
  Chronic pain intensity will be assessed at 3, 6, 9, and 12 months after surgery using A 0-10 numerical rating scale (0 means no pain and 10 means the worst pain)
morphine consumption | 48 hours after surgery
  Total morphine dose consumed during the second postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study
Access Criteria: The data will be available upon reasonable request from the corresponding author